CLINICAL TRIAL: NCT00957762
Title: Body Composition Assessment in Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: David R Gater MD, Ph D, Hunter Holmes McGuire VA
Other Study IDs: B6232I; HM12090
Record Dates: First submitted 2009-08-05; First posted 2009-08-12 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitus; Body Composition; Tetraplegia; Paraplegia; Spinal Cord Injury
Keywords: Body Composition; Glucose Tolerance; Insulin Sensitivity; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Quadriplegia; Paraplegia; Spinal Cord Injuries; Insulin Resistance; Metabolic Syndrome | interventions — Body Composition; Creb3l2 protein, rat

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Body Composition: 120 subjects will help create the regression models. The remaining 50 subjects will be recruited to determine if the equations work for the population.
  Interventions: Other: Body composition

INTERVENTIONS:
Other: Body composition — Day 1 testing will incorporate underwater weighing, Bod Pod, DXA, BIA and anthropometrics. Day 2 will include RMR, MRI, and testing at GCRC
  Other Names: Spinal Cord Injury; Percentage body fat

SUMMARY:
The purpose of this research is to evaluate different methods of measuring body composition (amount of fat, muscle, bone, and water in your body) and to determine relationships between body composition and other medical problems associated with spinal cord injury (SCI).

DETAILED DESCRIPTION:
A preliminary investigation in our laboratory has demonstrated the advantage of using 4-compartment modeling to assess body composition in SCI adults. In comparing body composition analyses techniques in 20 individuals with SCI, we found Total Error to be 8.0% with Dual X-ray Absorptiometry, 8.4% with hydrodensitometry, 11.5% with bioelectrical impedance analysis, and 21.8% with standard skinfold equations when compared to 4-compartment modeling, the currently accepted gold standard for body composition assessment. To date there is no gold standard for the determination of body composition in SCI individuals.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for participation will include men and women within the age range of 18-65 years old with C5-L2 Motor-Complete (ASIA A&B)
* SCI of duration greater than 12 months to ensure a homogenous sample.

Exclusion Criteria:

* Persons with uncompensated hypothyroidism, and/or renal disease will be excluded from the study.
* Additionally, individuals with uncontrolled autonomic dysreflexia, recent (within 3 months) deep vein thrombosis
* Pressure ulcers > Grade II will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a spinal cord injury of C5-L2 motor complete (AIS A&B only).
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To compare different methods of body composition analyses with the gold standard 4-compartment monitoring to determine accuracy and validity of those alternative, but less labor-intensive techniques. | 3 years

SECONDARY OUTCOMES:
To assess the relationship between % body fat, visceral fat, and markers of the metabolic syndrome, including Plasminogen Activator Inhibitor-1 (PAI-1), Thrombin-Activatable Fibrinolysis Inhibitor (TAFI), and high-sensitivity C-Reactive Protein (hsCRP) | 3 years
To develop body composition regression equations that can be easily utilized in a clinical setting to estimate risk for the metabolic syndrome in persons with SCI. | 3 years
To cross-validate the derived regression equations against the gold standard 4-compartment model in an independent group of persons with SCI. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David R Gater, MD, PhD, Principal Investigator — Hunter Holmes McGuire VAMC
Locations (1):
- Hunter Holmes McGuire Spinal Cord Injury Research Lab, Richmond, Virginia, United States